CLINICAL TRIAL: NCT05473988
Title: Optimization of Treatment Priority of the Manchester Triage System
Acronym: OPTIMTS
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OPTIMTS
Record Dates: First submitted 2022-07-12; First posted 2022-07-26 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Triage
MeSH Terms: interventions — Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Admission to General Ward Positive: Admission to General Ward Positive
  Interventions: Other: Admission to General Ward
- 30 Day Mortality Positive: 30 Day Mortality Positive
  Interventions: Other: 30 Day Mortality
- Admission to Intensive Care Unit Positive: Admission to Intensive Care Unit Positive
  Interventions: Other: Admission to Intensive Care Unit
- Admission to General Ward Negative: Admission to General Ward Negative
- 30 Day Mortality Negative: 30 Day Mortality Negative
- Admission to Intensive Care Unit Negative: Admission to Intensive Care Unit Negative

INTERVENTIONS:
Other: Admission to General Ward — Admission to General Ward
  Groups: Admission to General Ward Positive
Other: Admission to Intensive Care Unit — Admission to Intensive Care Unit
  Groups: Admission to Intensive Care Unit Positive
Other: 30 Day Mortality — 30 Day Mortality
  Groups: 30 Day Mortality Positive

SUMMARY:
In the emergency department, the urgency for treating patients is determined according to the Manchester Triage System. The parameters collected in this process are deterministically translated into a treatment priority.

The Manchester Triage System (MTS), which has been in use for at least 20 years, is a widely used, validated and standardized procedure for initial assessment in the emergency department - this initial assessment (triage) is done to prioritize medical assistance at a central point. Especially in emergency situations, critically endangered patients often require the deployment of a large part of the available staff at the same time - the medically correct triage of patients according to objective criteria in order to enable an adequate allocation of the available resources at the right time is the main objective. In the optimal case, each patient is treated by medical professionals within the time frame that is adequate for his/her health condition.

Using artificial intelligence methods, it may be possible to increase the accuracy of treatment priority assignment. In the best case, incorrect prioritization of patients can be prevented and medical care can be ensured for those patients who actually need it most urgently.

However, initial assessment, even if standardized and validated, still runs under limited resource conditions - time, space, material and personnel. Last but not least, the very idea of conducting an initial assessment limits its validity, and the results of the allocation fluctuate according to current research, although the determinants of this are currently unknown.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients that were triaged at the emergency department at the Kepler University Hospital in the period between 2015-12-01 to 2020-08-31.

Exclusion Criteria:

* None.

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: As described in the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 77976 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
AUROC for Classification of Admission to General Ward | 2015-12-01 to 2020-08-31
  AUROC for Classification of Admission to General Ward
AUROC for Classification of Admission to Intensive Care Unit | 2015-12-01 to 2020-08-31
  AUROC for Classification of Admission to Intensive Care Unit
AUROC for Classification of 30 Day Mortality | 2015-12-01 to 2020-08-31
  AUROC for Classification of 30 Day Mortality

SECONDARY OUTCOMES:
Confusion Matrix | 2015-12-01 to 2020-08-31
  Confusion Matrix Results: true positives, true negatives, false positive, false negatives and values calculated from these results.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tschoellitsch, MD, Principal Investigator — Kepler University Hospital and Johannes Kepler University, Linz, Austria
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No